CLINICAL TRIAL: NCT03919968
Title: Effect of Muay Thai vs. Circuit Training on the Health of Elderly: A Randomized Clinical Trial
Brief Title: Effect of Muay Thai vs. Circuit Training on the Cardiovascular Health of Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Bruna Thamyres Ciccotti Saraiva, Principal Investigator, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 91923318.7.0000.5402
Record Dates: First submitted 2019-03-19; First posted 2019-04-18 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Elderly
Keywords: Elderly; Martial Arts; Functional Training; Cardiovascular; Health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Martial Arts (Experimental): The training will be performed 3 times a week, for 12 weeks, during 60 minutes, being that will be divided into 20 min of general exercises, 20 min of specific exercises and 20 min of fight simulation and / or play activities. The activities will be carried out in a way adapted for the elderly. Will be used kickers, gauntlets, thorax and head protectors, shin guards, gloves, and other devices.
  Interventions: Behavioral: Functional Training
- Functional Training (Active Comparator): The training will be performed 3 times a week, for 12 weeks, during 60 minutes, being that will be divided into 20 min of general exercises, 20 min of specific exercises and 20 min of play activities. The activities will be carried out in a way adapted for the elderly. Will be carried out neuromotor control / coordination, balance, flexibility and static and dynamic stabilization. They will also have acceleration and deceleration activities, rotation and counter-rotation, extension and counter-extension, flexion and counter-flexion.
  Interventions: Behavioral: Martial Arts

INTERVENTIONS:
Behavioral: Martial Arts — The training will be performed 3 times a week, for 12 weeks, during 60 minutes, being that will be divided into 20 min of general exercises, 20 min of specific exercises and 20 min of fight simulation and / or play activities. The activities will be carried out in a way adapted for the elderly. Will be used kickers, gauntlets, thorax and head protectors, shin guards, gloves, and other devices.
  Arms: Functional Training
Behavioral: Functional Training — The training will be performed 3 times a week, for 12 weeks, during 60 minutes, being that will be divided into 20 min of general exercises, 20 min of specific exercises and 20 min of play activities. The activities will be carried out in a way adapted for the elderly. Will be carried out neuromotor control / coordination, balance, flexibility and static and dynamic stabilization. They will also have acceleration and deceleration activities, rotation and counter-rotation, extension and counter-extension, flexion and counter-flexion.
  Arms: Martial Arts

SUMMARY:
The elderly will be recruited, after meeting the inclusion criteria, will be submitted to data collection, all necessary assessments for the study and after 12 weeks, the same data will be collected, so that the elderly are self-control. After the second collection, the elderly will be randomized into two groups: the Muay Thai group and the functional training group. Both groups will train three times a week for 60 min and for 12 weeks. The training will be divided into 20 min of general exercises, 20 min of specific exercises and 20 min of fight simulation and/or play activities. At the end of the 12 weeks of intervention, evaluations and data collection will be performed again.

DETAILED DESCRIPTION:
Will be recruited through media resources at least 50 elderly people aged between 60 and 89 years.

Inclusion Criteria:

Being literate; Age between 60 and 89 years; Ability to perform moderate-intensity exercises determined by the American College Sports Medicine (ACSM) assessment questionnaire; Medical certificate stating that the elderly are able to exercise; Sign the informed consent form.

Exclusion Criteria:

Perform any other systematic practice of physical exercise, in addition to regular physical activity, such as walking; Present serious cardiovascular pathologies; Present serious neurological pathologies; Present use of crutches, walking sticks, walkers, wheelchairs or other similar utensils; Present self-report of locomotion difficulties to carry out the intervention practice.

These will have three moments of evaluations. Baseline, pre intervention (3 months) and post intervention (6 months) since the elderly will be controls themselves. They will perform anthropometric measurements, answer physical activity questionnaires, sedentary behavior, sleep quality, anxiety and depression, quality of life, cognition evaluation, body composition measurements, functional capacity, autonomic cardiac modulation, hemodynamics, flow and thickness of arteries, as well as flow-mediated dilatation. After the second-step measures (pre intervention 3 months), they will be randomized into two groups: Muay Thai and functional training. The functional training will be performed 3 times a week, for 12 weeks, during 60 minutes, being that will be divided into 20 min of general exercises, 20 min of specific exercises and 20 min of play activities. The activities will be carried out in a way adapted for the elderly. Will be carried out neuromotor control / coordination, balance, flexibility and static and dynamic stabilization. They will also have acceleration and deceleration activities, rotation and counter-rotation, extension and counter-extension, flexion and counter-flexion. The Muay Thai training will be performed 3 times a week, for 12 weeks, during 60 minutes, being that will be divided into 20 min of general exercises, 20 min of specific exercises (punches, kicks, knees, elbows, defenses and dodges) and 20 min of fight simulation and / or play activities. The activities will be carried out in a way adapted for the elderly. Will be used kickers, gauntlets, thorax and head protectors, shin guards, gloves, and other devices.

ELIGIBILITY:
Inclusion Criteria:

* Being literate;
* Age between 60 and 89 years;
* Ability to perform moderate-intensity exercises determined by the American College Sports Medicine (ACSM) assessment questionnaire;
* Medical certificate stating that the elderly are able to exercise;
* Sign the informed consent form.

Exclusion Criteria:

* Perform any other systematic practice of physical exercise, in addition to regular physical activity, such as walking;
* Present serious cardiovascular pathologies;
* Present serious neurological pathologies;
* Present use of crutches, walking sticks, walkers, wheelchairs or other similar utensils;
* Present self-report of locomotion difficulties to carry out the intervention practice.

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Autonomic Cardiac Modulation | Change from Baseline Autonomic Cardiac Modulation to 3 months after intervention
  The heart rate variability will be collected by means of the POLAR V800.

SECONDARY OUTCOMES:
Physical activity level - objective measure | Pre baseline, Post 3 months (Pre-intervention) and Post 6 months (Post-intervention)
  Will be collected 7 days of accelerometry by ActiGraph's triaxial accelerometer wGT3X-BT giving the measure in counts per minute.
Self-reported physical activity level questionnaire | Pre baseline, Post 3 months (Pre-intervention) and Post 6 months (Post-intervention)
  The modified Baecke's questionnaire for the elderly will be used to evaluate the practice of physical activity and a score will be calculated, both for total practice and for domains, the quartile of the evaluated elderly will be calculated and below 25 will be considered insufficiently active, above with sufficient physical activity practice
Self-reported sedentary behaviour questionnaire | Pre baseline, Post 3 months (Pre-intervention) and Post 6 months (Post-intervention)
  The participants were asked to state the total time they usually spent (expressed in minutes per day) sitting or reclining including at work, at home, getting to and from places, or with friends (e.g. sitting at a desk, sitting with friends, travelling in car, bus, train, reading, playing cards or watching television).
Quality of life questionnaire | Pre baseline, Post 3 months (Pre-intervention) and Post 6 months (Post-intervention)
  The questionnaire validated for the elderly will be applied the Short Form Health Survey (SF-36), composed of 36 questions with a score ranging from 0 to 100, being 0 the worst and 100 best.
Force- objective measure | Pre baseline, Post 3 months (Pre-intervention), Post-intervention 6 months
  Will be performed the American Alliance for Health, Physical Education, Recreation and Dance (AAHPERD) battery tests. Will use a 2-kg halter to measure upper limb strength, make as many elbow push-ups with the halter on hand in 30 seconds the final test result is the best performance of two trials performed. Below 7 repetitions is considered weak strength, above is good.
Flexibility- objective measure | Pre baseline, Post 3 months (Pre-intervention) and Post 6 months (Post-intervention)
  Will be performed the American Alliance for Health, Physical Education, Recreation and Dance (AAHPERD) battery tests. Will be by means of sitting and reaching adapted. Below 47 cm is considered weak flexibility, above is good.
Agility and dynamic balance - objective measure | Pre baseline, Post 3 months (Pre-intervention) and Post 6 months (Post-intervention)
  Will be performed the American Alliance for Health, Physical Education, Recreation and Dance (AAHPERD) battery tests. It will be evaluated sitting in a chair with two cones positioned one on the right side and another on the left the goal is to turn the cones and sit and time will be timed. Two attempts are made and the shortest time is counted in seconds as the final result.
Cardiorespiratory capacity- 6-minute walk test | Pre baseline, Post 3 months (Pre-intervention) and Post 6 months (Post-intervention)
  The teste will be performed in a 30-meter corridor, and the subjects were instructed to keep walking for 6 minutes. The best way will be considered for analysis. Below 400-meter is considered with low cardiorespiratory capacity, above is good.
Bone Mineral Density | Pre baseline, Post 3 months (Pre-intervention) and Post 6 months (Post-intervention)
  The bone mineral density will be evaluated through dual energy x-ray absorptiometry.
Body fat | Pre baseline, Post 3 months (Pre-intervention) and Post 6 months (Post-intervention)
  The body fat will be evaluated using the octopolar apparatus InBody 720 (Copyright®, 1996-2006, by Biospace Corporation, USA) in percentage.
Fat mass | Pre baseline, Post 3 months (Pre-intervention) and Post 6 months (Post-intervention)
  The fat mass will be evaluated using the octopolar apparatus InBody 720 (Copyright®, 1996-2006, by Biospace Corporation, USA) in kilograms.
Muscle mass | Pre baseline, Post 3 months (Pre-intervention) and Post 6 months (Post-intervention)
  The muscle mass will be evaluated using the octopolar apparatus InBody 720 (Copyright®, 1996-2006, by Biospace Corporation, USA) in kilograms.
Cognitive ability | Pre baseline, Post 3 months (Pre-intervention) and Post 6 months (Post-intervention)
  The cognitive capacity of the elderly will be evaluated by the Mini-mental state exam. Consists of two parts, one that includes guidance, memory and attention, with a maximum score of 21 points, and another that addresses specific skills such as naming and comprehension, with a maximum score of 9 points, totaling a score of 30 points. Higher scores indicate greater cognitive performance.
Systolic Blood pressure | Pre baseline, Post 3 months (Pre-intervention) and Post 6 months (Post-intervention)
  The systolic blood pressure will be measured by means of the omron digital oscillometric device.
Diastolic Blood pressure | Pre baseline, Post 3 months (Pre-intervention) and Post 6 months (Post-intervention)
  The diastolic blood pressure will be measured by means of the omron digital oscillometric device.
Resting heart rate | Pre baseline, Post 3 months (Pre-intervention) and Post 6 months (Post-intervention)
  The resting heart rate will be measured by means of the omron digital oscillometric device.
Blood flow of the arteries | Pre baseline, Post 3 months (Pre-intervention) and Post 6 months (Post-intervention)
  To verify the blood flow of the carotid and femoral arteries will be used the ultrasound doopler
Thickness of the arteries | Pre baseline, Post 3 months (Pre-intervention) and Post 6 months (Post-intervention)
  To verify the thickness of the carotid and femoral arteries will be used the ultrasound doopler
Flow-mediated dilation | Pre baseline, Post 3 months (Pre-intervention) and Post 6 months (Post-intervention)
  Flow-mediated dilation will be assessed by pre and post occlusion doopler ultrasound of the brachial artery.
Anxiety and depression questionnaire | Pre baseline, Post 3 months (Pre-intervention) and Post 6 months (Post-intervention)
  Will be assessed by hospital anxiety and depression scale aims to detect mild degrees of affective disorders in non-psychiatric settings. It consists of 14 multiple choice items, seven of which are for anxiety assessment and seven for depression. Each item can be punctuated from 0 to 3, reaching a maximum of 21 points in each subscale. An indicative score of anxiety equal to or greater than 8; and a score indicative of depression equal to or greater than 9.

CONTACTS AND LOCATIONS:
Overall Officials: Diego Christofaro, PhD, Principal Investigator — Universidade Estadual Paulista - UNESP
Locations (1):
- Bruna T C Saraiva, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saraiva BTC, Franchini E, Ribeiro AS, Gobbo LA, Correia MA, Vanderlei LCM, Ferrari G, Tebar WR, Christofaro DGD. Effects of 12 weeks of functional training vs. Muay Thai on cardiac autonomic modulation and hemodynamic parameters in older adults: a randomized clinical trial. BMC Cardiovasc Disord. 2024 Aug 17;24(1):433. doi: 10.1186/s12872-024-04096-3. PMID 39153977